CLINICAL TRIAL: NCT05424341
Title: Comparative Effects Of Muscle Energy Technique And Counter Strain Technique On Pain, Functional Status And Satisfaction Level In Planter Fasciitis Patients
Brief Title: Effects Of Muscle Energy Versus Counter Strain Technique on Pain, Function and Satisfaction Level in Planter Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Ayesha Jamil, Assistant Professor, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Taliah Bashir Sindhu
Record Dates: First submitted 2022-06-08; First posted 2022-06-21 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Plantar Fasciitis
Keywords: Counterstrain, Function, METs, Pain, Plantar Fasciitis, Satisfaction
MeSH Terms: conditions — Fasciitis, Plantar; Pain; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Group A: Muscle energy technique along with routine physical therapy, Group B: Counterstrain technique along with routine physical therapy
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): This group will receive muscle energy technique along with routine physical therapy. This protocol will be given for 3 alternative days for 2 weeks . Each session will be of 50 mins. Data will be collected at baseline , at 1st week and at 2nd week.
  Interventions: Other: Muscle Energy Technique
- Group B (Active Comparator): This group will receive counterstrain technique along with routine physical therapy. This protocol will be given for 3 alternative days for 2 weeks . Each session will be of 50 mins. Data will be collected at baseline , at 1st week and at 2nd week.
  Interventions: Other: Counterstrain Technique

INTERVENTIONS:
Other: Muscle Energy Technique — For Gastrocnemius muscle, subject will be in supine position keeping knee fully extended and therapist on affected side in walking position. The subject's ankle joint will be dorsiflexed until a resistance feel and will ask to hold this position and exert 20% of force towards plantar flexion for a period of 5 to 7 seconds. Resistance will be released and relaxation of 5 seconds will be given during which the ankle will was passively dorsiflexed to a new barrier. 5 repetitions will be given.
  Arms: Group A
Other: Counterstrain Technique — Therapist places thumb on tender point at plantar fascia insertion while patient in supine position with ipsilateral knee flexed. Plantar flex the toes and ankle while monitoring sore site with thumb, curling around tender point until monitoring thumb feels symptomatic relief. Supination/pronation of foot will be added if necessary. The position of ease will be maintained for 90 secs until tissues beneath monitoring thumb softens. Tender spot is re-evaluated once the foot is returned to neutral without moving the thumb. It will be repeated 3 times for 30 secs resting interval in-between
  Other Names: Spontaneous Release by Positioning
  Arms: Group B

SUMMARY:
Previous studies has discussed the effects of muscle energy technique and counterstrain technique in upper trapezius and low back pain but no comparative study is found on planter fasciitis patients. In this study we are going to compare the effects of muscle energy technique and counterstrain technique with routine physical therapy in relation with pain, functional status and satisfaction level in planter fasciitis patients

DETAILED DESCRIPTION:
Heel pain is one of the most prevalent musculoskeletal diseases of the lower limb, affecting both physically active and sedentary people. Amongst the possible causes, planter fasciitis is one of the most common cause of heel pain.

Planter fasciitis is a degenerative syndrome resulting from the repeated injury at its origin on the calcaneus. Its most common symptom is discomfort in the plantar area of the foot and, more specifically, in the inferior part of the heel. It is frequently more intense while taking your first steps in the morning or after a period of physical inactivity, and it worsens with prolonged standing or weight-lifting activities. It is not frequently linked to nocturnal discomfort or paresthesia.

Different physiotherapy treatment conventions help in pain relieving for example, rest, taping, stretching, orthosis-night brace, Silicon heel cups and myofascial release. This study will compare the effects of Muscle Energy Technique versus Counterstrain Technique in patients with plantar Fasciitis.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 68 years.

  * Both male and female.
  * Patients are clinical diagnosed by the orthopedic surgeon.
  * Patients present with pain that persist for more than 4 weeks in heel and planter surface of foot.
  * Pain with the first steps after inactivity

Exclusion Criteria:

* • Patients with history of ankle and foot fracture.

  * Congenital or acquired deformity of ankle and foot.
  * Patients with arthritis.
  * Pervious history of surgery for planter fasciitis.
  * Patients use an assistive device for walking.
  * Patients use corticosteroid injection in heel.

Ages: 20 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Change in pain intensity will be measured at baseline, at end of first week, at end of second week
  Pain intensity will be measured by Visual Analogue Scale (VAS)
Function | Change in Functional Status will be measured at baseline, at end of first week, at end of second week
  Functional status will be measured by Foot and Ankle Ability Measure (FAAM)
Satisfaction Level | Level of satisfaction will be observed at end of First Session, at end of first week, at end of second week
  Satisfaction level will be measured by Short-Form Patient Satisfaction Questionnaire (PSQ-18)

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Jamil, M.Phil, Study Chair — University of Lahore
Locations (1):
- The University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Immediately after publication
Time Frame: Beginning 9 months and ending on 36th month